CLINICAL TRIAL: NCT07215689
Title: A Prospective, Randomized, Double-Blind, Placebo Controlled Clinical Study to Evaluate the Effects of KSM- 66 Ashwagandha® Capsule (300 mg) on Skin and Hair Health in Healthy Men and Women
Brief Title: Effects of KSM-66 Ashwagandha® (300 mg) on Skin and Hair Health in Healthy Men and Women"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ixoreal-HS-CT-05-22
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Skin Health; Hair Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1: Interventional KSM-66 Ashwagandha® capsule (300 mg) (Active Comparator): KSM-66 Ashwagandha® capsule (300 mg) orally twice daily after food with a glass of water or milk for 90 ± 4 days.
  Interventions: Dietary Supplement: KSM-66 Ashwagandha® capsule
- Treatment Arm 2: Identical placebo capsule (Placebo Comparator): Placebo capsule containing starch (300 mg) orally twice daily after food with a glass of water or milk for 90 ± 4 days.
  Interventions: Other: Placebo Capsule(s)

INTERVENTIONS:
Dietary Supplement: KSM-66 Ashwagandha® capsule — Single off-white capsule contains 300mg Ashwagandha root extract powder only
  Arms: Treatment Arm 1: Interventional KSM-66 Ashwagandha® capsule (300 mg)
Other: Placebo Capsule(s) — Single off-white capsule contains starch powder only
  Arms: Treatment Arm 2: Identical placebo capsule

SUMMARY:
Hair and skin play major roles in protecting the body, and maintaining their health is essential. Poor hair and skin health have become increasingly common due to the stress associated with modern lifestyles. Effective and time-efficient treatments for hair and skin health remain limited. Although hair loss, baldness, and skin issues are not life-threatening, managing these conditions is important because of the psychological and social complications-such as anxiety and depression-they can cause. There is an unmet need for therapies that provide safe and long-term improvements in hair and skin health.

Many individuals seek Complementary and Alternative Medicine (CAM) to identify natural and effective options for these conditions. Adaptogens such as Ashwagandha (Withania somnifera) have long been studied for their potential to reduce stress and modulate cortisol levels in the body. Reducing stress may help prevent inflammation, a common contributor to hair shedding and loss. Ashwagandha also contains antioxidants and amino acids that may strengthen the hair and minimize breakage. Traditionally, Ashwagandha has been recognized for its multiple health benefits, including support for hair and skin wellness. However, there remains limited scientific evidence to substantiate these traditional claims, underscoring the need for controlled clinical evaluation.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical study is designed to evaluate the effects of KSM-66 Ashwagandha® (300 mg capsule) on hair and skin health in healthy men and women. The study aims to assess whether Ashwagandha supplementation can improve parameters related to skin hydration, elasticity, and barrier function, as well as hair density and strength.

Participants will be randomized to receive either KSM-66 Ashwagandha or placebo for the study duration. The assessments will include validated questionnaires, dermatological evaluations, and instrumental measurements of skin and hair parameters. The results are expected to provide evidence on the potential efficacy and safety of Ashwagandha in supporting hair and skin health through its adaptogenic and stress-modulating properties.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women participants ≥ 18 years and ≤60 years of age.
2. Willingness to follow the protocol requirements as evidenced by written informed consent.
3. Participants who were on consistent dietary, hair, and skin product 3 months prior to start of the study and are willing to follow the same during the study.
4. Participants who agree not to use any medication (prescription and over the counter), including vitamins and minerals, during or before the course of this study.
5. Participants with mild to moderate hair loss classified as the Norwood-Hamilton type II, III, IV and V in males and Ludwig type I and II in females.
6. Willing to come for all follow-up visits.
7. Participants who agree not to cut hair for the entire duration of the study.
8. Participants willing to undergo Trichoscan evaluation and not to wash their hair 48 hours before the visit.
9. Participants or LAR can and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements.
10. Participants who agree to take investigational product (i.e., Till Day 90 ± 4 ± 4).

Exclusion Criteria:

1. Participants having any clinically significant medical history, medical finding including rosacea, eczema, psoriasis, and atopic dermatitis or an on-going medical or psychiatric condition exists which in the opinion of the Investigator could jeopardize the safety of the subject, impact validity of the study results or interfere with the completion of study according to the protocol.
2. Participants on any medication or supplement for hair loss, including finasteride, any other 5 α-reductase inhibitor, minoxidil, steroids, or hormonal products, during the 3 months prior to study commencement.
3. Participants having a history of hypersensitivity reactions (i.e., allergic or oversensitivity to study medication).
4. Participants who have undergone or plan to undergo hair transplantation surgery during the study period.
5. Participants with facial skin cancer.
6. Participants with sunburn, moderate to pronounced suntan, uneven skin tones, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results.
7. Participants with severe seborrheic dermatitis, alopecic disease, except for androgenic alopecia, and scalp disorders, such as scalp psoriasis and infection.
8. Participants who have participated in a clinical study during the preceding 180 days.
9. Participants having eating disorders (i.e., bulimia, psychogenic eating disorders, etc.).
10. Pregnant and lactating females
11. Participants with alcohol addiction or persistent abuse of drugs of dependence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of KSM-66 Ashwagandha formulation on skin health in adult healthy men and women, in terms of TEWL (Trans Epidermal Water Loss) | Baseline, Week 12
  Mean change in TEWL from Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1) to Visit 3, End of study (Week 12)

SECONDARY OUTCOMES:
Change in Hair Density (n/cm²) | Baseline, Week 12
  To evaluate the effect of KSM-66 Ashwagandha on hair density from Baseline (Day 1) to Week 12 using Trichoscan analysis.
To evaluate the efficacy of KSM-66 Ashwagandha formulation on skin health in terms of QoL for Skin using the Dermatology Life Quality Index (DLQI). | Baseline, Week 12
  To evaluate the efficacy of KSM-66 Ashwagandha formulation on skin health in terms of quality of life using the Dermatology Life Quality Index (DLQI) questionnaire.
  Measurement Scale:
  DLQI total score ranges from 0 to 30, where
  0-1: No effect on patient's life,
  2-5: Small effect,
  6-10: Moderate effect,
  11-20: Very large effect,
  21-30: Extremely large effect. Lower scores indicate better dermatological quality of life (i.e., improvement).
To evaluate the efficacy of KSM-66 Ashwagandha formulation on hair in terms of QoL for Hair using the Hair Skindex-29 Questionnaire | Baseline, Week 12
  To evaluate the efficacy of KSM-66 Ashwagandha formulation on hair health using the Hair Skindex-29 Questionnaire.
  Measurement Scale:
  The Hair Skindex-29 is a validated 29-item questionnaire assessing the effects of hair conditions on quality of life, with a total score range of 0-100.
  Higher scores represent worse quality of life, while lower scores indicate improvement.
To evaluate the effects of KSM-66 Ashwagandha formulation on hair and skin in terms of self-assessment for skin and hair health | Baseline, Week 12
  To evaluate the participant's perceived improvement in hair and skin health using a 5-point Likert scale.
  Measurement Scale:
  Scores range from 1 to 5, where
  1. = Very much worse,
  2. = Worse,
  3. = No change,
  4. = Improved,
  5. = Very much improved. Higher scores indicate better improvement as perceived by the participant.
To evaluate the effects of KSM-66 Ashwagandha formulation on hair and skin in terms of physician's global assessment | Baseline, Week 12
  To evaluate the investigator's overall assessment of improvement in hair and skin health using the Global Physician Assessment scale.
  Measurement Scale:
  A 5-point Likert scale, where
  1. = Very much worse,
  2. = Worse,
  3. = No change,
  4. = Improved,
  5. = Very much improved. Higher scores indicate better improvement as assessed by the physician.
Change in Hair Diameter (µm) | Baseline, Week 12
  To evaluate the effect of KSM-66 Ashwagandha on mean hair diameter from Baseline (Day 1) to Week 12 using Trichoscan analysis.
To evaluate the safety of KSM-66 Ashwagandha formulation in healthy men and women | Baseline, Week 12
  Number and proportion of Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Event (TESAE)
Change in Hair Growth Rate (mm/day) | Baseline, Week 12
  To assess the change in average hair growth rate from Baseline (Day 1) to Week 12 using Trichoscan analysis.
Change in Anagen/Telogen Ratio | Baseline, Week 12
  To evaluate changes in the Anagen/Telogen ratio as an indicator of hair growth phase balance from Baseline (Day 1) to Week 12 using Trichoscan analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No